CLINICAL TRIAL: NCT01984229
Title: An Open-Label, Three-Period, Fixed Sequence Study to Investigate the Effect of Multiple Oral Doses of Posaconazole, a Potent Cytochrome P450 3A Inhibitor, on the Single Dose Pharmacokinetics of RO5424802 in Healthy Subjects
Brief Title: A Study of the Effects of Posaconazole on Alectinib (RO5424802) Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP28990
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — alectinib; posaconazole

ARMS (2):
- Cohort A (Experimental): There will be 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 14), and Period 3 (Days 15 to 18). Alectinib will be administered as a 40 milligrams (mg) single oral dose on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants). On Days 8 to 14 (Period 2) and Days 15 to 18 (Period 3) posaconazole will be administered as a 400-mg twice daily (BID) oral dose after a high-fat meal. The follow-up assessments will occur within 10 to 14 days after the last dose of posaconazole.
  Interventions: Drug: Alectinib; Drug: Posaconazole
- Cohort B (Experimental): There will be 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 14), and Period 3 (Days 15 to 21). Alectinib will be administered as a single oral dose at the dose selected based on Cohort A data on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants). On Days 8 to 14 (Period 2) and Days 15 to 21 (Period 3) posaconazole will be administered as a 400-mg BID oral dose after a high-fat meal. The follow-up assessments will occur within 10 to 14 days after the last dose of posaconazole.
  Interventions: Drug: Alectinib; Drug: Posaconazole

INTERVENTIONS:
Drug: Alectinib — Alectinib will be administered as a single oral dose on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants).
  Other Names: RO5424802
Drug: Posaconazole — Posaconazole will be administered as a 400-mg BID oral dose after a high-fat meal on Days 8 to 14 (Period 2) and Days 15 to 18 or 21 (Period 3).

SUMMARY:
This open-label study will investigate whether multiple oral doses of posaconazole affect the single dose pharmacokinetics of alectinib in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 to 32 kilogram per square meter (kg/m^2)
* Male volunteers must use effective contraception as outlined in the protocol
* Willingness to abstain from alcohol and xanthine-containing beverages or food (coffee, tea, cola, chocolate and "energy drinks") from 72 hours prior to the first dose until discharged
* Willingness to avoid prolonged sun exposure and guard against sunburn during study and follow-up

Exclusion Criteria:

* Clinically significant medical history or findings in physical examination, vital signs, or laboratory test results prior to study start
* Positive screening tests for hepatitis B or C, human immunodeficiency virus (HIV), alcohol, drugs of abuse, or tobacco
* Women of childbearing potential, or males with pregnant or lactating partners
* Regular smoking within 6 months prior to first dosing. Participants should avoid smoky environments for at least 1 week prior to each cotinine screen
* Excessive alcohol consumption
* Use of any metabolic inducers (including herbals such as St. John's Wort) within 4 weeks or 5 half-lives (whichever is longer) before the first dose of study medication, including but not limited to: rifampin, rifabutin, glucocorticoids, carbamazepine, phenytoin and phenobarbital
* Strenuous activity, sunbathing, or contact sports are not allowed from 4 days prior to entry into the clinical site until study follow-up
* Participation in an investigational drug or device study within 45 days (or 6 months for biologic therapies) prior to first dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole: There were 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 14), and Period 3 (Days 15 to 18). Alectinib was administered as a 40 milligrams (mg) single oral dose on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants). On Days 8 to 14 (Period 2) and Days 15 to 18 (Period 3) posaconazole was administered as a 400-mg twice daily (BID) oral dose after a high-fat meal. The follow-up assessments occurred within 10 to 14 days after the last dose of posaconazole.
- Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole: There were 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 14), and Period 3 (Days 15 to 21). Alectinib was administered as a 300-mg single oral dose on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants). On Days 8 to 14 (Period 2) and Days 15 to 21 (Period 3) posaconazole was administered as a 400-mg BID oral dose after a high-fat meal. The follow-up assessments occurred within 10 to 14 days after the last dose of posaconazole.
Period: Period 1
Arm/Group | Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole | Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole | Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole | Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0
Period: Safety Follow-up Period
Arm/Group | Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole | Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole
Started | 6 | 17
Completed | 4 | 16
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all participants who received at least 1 dose of study drug and had at least 1 after dosing safety assessment.
Groups:
- Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole: There were 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 14), and Period 3 (Days 15 to 18). Alectinib was administered as a 40-mg single oral dose on Day 1 (Period 1) and Day 15 (Period 3) with an identical standardized meal (identical meal on Day 1 and Day 15 across all participants). On Days 8 to 14 (Period 2) and Days 15 to 18 (Period 3) posaconazole was administered as a 400-mg BID oral dose after a high-fat meal. The follow-up assessments occurred within 10 to 14 days after the last dose of posaconazole.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Alectinib 40mg, Posaconazole, Alectinib+Posaconazole | Cohort B:Alectinib 300mg, Posaconazole, Alectinib+Posaconazole | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.50) | 38.5 (8.40) | 38.3 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 15 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Alectinib: Cohort A
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: Pharmacokinetic (PK) Analysis Population [Cohort A] consisted of all participants who received both scheduled doses of Alectinib, and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Cohort A: Alectinib (Period 1): Alectinib was administered as a 40-mg single oral dose on Day 1 (Period 1).
- Cohort A: Alectinib + Posaconazole (Period 3): Alectinib was administered as a 40-mg single oral dose on Day 15 (Period 3). On Days 15 to 18 (Period 3) posaconazole was administered as a 400-mg BID oral dose after a high-fat meal.
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
nanograms per milliliter (ng/mL) | 27.6 (6.61) | 35.0 (10.8)

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Alectinib: Cohort A
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Cohort A]
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
hours*nanograms per milliliter (h*ng/mL) | 634 (133) | 1030 (270)

3. Primary Outcome: Cmax of Alectinib: Cohort B
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period, and additional samples were collected in Period 3 at 120, 144, 168, 192, and 216 hours after dosing
Population: PK Analysis Population [Cohort B] consisted of all participants who received both scheduled doses of Alectinib, and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort B: Alectinib (Period 1): Alectinib was administered as a 300-mg single oral dose on Day 1 (Period 1).
- Cohort B: Alectinib + Posaconazole (Period 3): Alectinib was administered as a 300-mg single oral dose on Day 15 (Period 3). On Days 15 to 21 (Period 3) posaconazole was administered as a 400-mg BID oral dose after a high-fat meal.
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
ng/mL | 147 (39.3) | 171 (38.2)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); Analysis of variance (ANOVA) was applied to the log-transformed PK parameter and then back transformed to provide geometric least square mean ratios (Period 3/Period 1) and confidence intervals (CIs); Test type: Superiority or Other; Geometric Least Square Mean Ratio = 118, 90% CI 2-sided [102 to 137] — The reported values are percentages of geometric least square mean ratio

4. Primary Outcome: AUClast of Alectinib: Cohort B
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
h*ng/mL | 2770 (545) | 4910 (893)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); ANOVA was applied to the log-transformed PK parameter and then back transformed to provide geometric least square mean ratios (Period 3/Period 1) and CIs; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 177, 90% CI 2-sided [159 to 198] — The reported values are percentages of geometric least square mean ratio

5. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of RO5424802: Cohort B
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
h*ng/mL | 2850 (549) | 4990 (888)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 175, 90% CI 2-sided [157 to 195] — The reported values are percentages of geometric least square mean ratio

6. Secondary Outcome: Cmax of RO5468924: Cohort A
Description: RO5468924 is M4 metabolite of Alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Cohort A]
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
ng/mL | 6.52 (1.59) | 2.54 (0.296)

7. Secondary Outcome: AUClast of RO5468924: Cohort A
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). RO5468924 is M4 metabolite of Alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Cohort A]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
h*ng/mL | 138 (36.8) | 65.1 (20.4)

8. Secondary Outcome: AUC0-inf of RO5468924: Cohort A
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf). RO5468924 is M4 metabolite of Alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Cohort A]. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 3
h*ng/mL | 201 (35.9) | 256 (94.5)

9. Secondary Outcome: Cmax of RO5468924: Cohort B
Description: RO5468924 is M4 metabolite of Alectinib.
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
ng/mL | 59.6 (27.1) | 15.5 (4.0)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 28.7, 90% CI 2-sided [23.1 to 35.5] — The reported values are percentages of geometric least square mean ratio

10. Secondary Outcome: AUClast of RO5468924: Cohort B
Description: as for outcome 7
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
h*ng/mL | 1460 (562) | 910 (211)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 66.2, 90% CI 2-sided [56.7 to 77.4] — The reported values are percentages of geometric least square mean ratio

11. Secondary Outcome: AUC0-inf of RO5468924: Cohort B
Description: as for outcome 8
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
h*ng/mL | 1550 (569) | 1110 (284)
Statistical Analysis 1: Comparison: Cohort B: Alectinib (Period 1) vs Cohort B: Alectinib + Posaconazole (Period 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 75.1, 90% CI 2-sided [64.4 to 87.7] — The reported values are percentages of geometric least square mean ratio

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alectinib: Cohort A
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK analysis population [Cohort A]
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
hours | 8.15 [6.00 to 12.0] | 8.00 [4.00 to 11.9]

13. Secondary Outcome: Tmax of Alectinib: Cohort B
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Cohort B]
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
hours | 8.00 [6.00 to 12.0] | 8.00 [6.00 to 11.9]

14. Secondary Outcome: Tmax of RO5468924: Cohort A
Description: RO5468924 is M4 metabolite of Alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK analysis population [Cohort A]
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
hours | 12.0 [6.03 to 12.0] | 11.9 [6.00 to 11.9]

15. Secondary Outcome: Tmax of RO5468924: Cohort B
Description: RO5468924 is M4 metabolite of Alectinib.
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
hours | 12.0 [6.00 to 12.0] | 11.9 [6.00 to 12.0]

16. Secondary Outcome: Metabolite/Parent Ratio for AUC0-inf: Cohort B
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf). RO5468924 is M4 metabolite of Alectinib. The ratio is molecular weight adjusted.
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
ratio | 0.541 (0.12) | 0.232 (0.02)

17. Secondary Outcome: Metabolite/Parent Ratio for Cmax: Cohort B
Description: RO5468924 is M4 metabolite of Alectinib. The ratio is molecular weight adjusted.
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
ratio | 0.393 (0.10) | 0.0953 (0.01)

18. Secondary Outcome: Terminal Half-life (t1/2) of Alectinib: Cohort A
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK analysis population [Cohort A]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 5
hours | 19.6 (2.37) | 26.9 (3.22)

19. Secondary Outcome: t1/2 of Alectinib: Cohort B
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
hours | 18.4 (4.36) | 24.8 (5.08)

20. Secondary Outcome: t1/2 of RO5468924: Cohort A
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. RO5468924 is M4 metabolite of Alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 5 | 3
hours | 23.9 (9.92) | 79.6 (47.2)

21. Secondary Outcome: t1/2 of RO5468924: Cohort B
Description: as for outcome 20
Time Frame: as for outcome 3
Population: PK Analysis Population [Cohort B]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort B: Alectinib (Period 1) | Cohort B: Alectinib + Posaconazole (Period 3)
Number analyzed (Participants) | 16 | 16
hours | 25.3 (4.12) | 69.6 (22.7)

ADVERSE EVENTS:
Time Frame: Day 1 up to 10 to 14 days after last dose of posaconazole (Cohort A: maximum up to 28 to 32 days; Cohort B: maximum up to 31 to 35 days)
Description: Safety Analysis Set. Only 5 participants were evaluable for adverse events in Cohort A: Alectinib + Posaconazole (Period 3) arm.
Groups:
- Cohort A: Posaconazole (Period 2); Cohort B: Posaconazole (Period 2): Posaconazole was administered as a 400-mg BID oral dose on Days 8 to 14 (Period 2) after a high-fat meal.
Arm/Group | Cohort A: Alectinib (Period 1) | Cohort A: Posaconazole (Period 2) | Cohort A: Alectinib + Posaconazole (Period 3) | Cohort B: Alectinib (Period 1) | Cohort B: Posaconazole (Period 2) | Cohort B: Alectinib + Posaconazole (Period 3)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/6 | 3/6 | 2/5 | 3/17 | 4/17 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Alectinib (Period 1) (N=6) | Cohort A: Posaconazole (Period 2) (N=6) | Cohort A: Alectinib + Posaconazole (Period 3) (N=5) | Cohort B: Alectinib (Period 1) (N=17) | Cohort B: Posaconazole (Period 2) (N=17) | Cohort B: Alectinib + Posaconazole (Period 3) (N=17)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.